CLINICAL TRIAL: NCT02673905
Title: Randomized, Multi-center Phase II Clinical Trial for the Regeneration of Cartilage Lesions in the Knee Using Nasal Chondrocyte-based Tissue (N-TEC) or Nasal Chondrocyte-based Cell (N-CAM)-Therapies
Brief Title: Clinical Trial for the Regeneration of Cartilage Lesions in the Knee
Acronym: NosetoKnee2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University Hospital Freiburg (Other); I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other); General Hospital Sveti Duh (Other); Fraunhofer-Institut für Silicatforschung ISC (Unknown); Orthopaedische Klinik Koenig-Ludwig-Haus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NosetoKnee2
Record Dates: First submitted 2016-02-01; First posted 2016-02-04 (Estimated); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Tear; Knee, Cartilage, Articular
Keywords: nasal chondrocytes; articular chondral lesions; tissue engineering; femoral condyle; trochlea
MeSH Terms: conditions — Lacerations | interventions — Histocompatibility Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- N-TEC (tissue engineered product) (Experimental): N-TEC is based on autologous nasal chondrocytes expanded and further cultured on type I/III collagen membrane for 2 weeks to allow the cells to produce extracellular matrix containing cartilage specific Proteins. The IMP is implanted in the knee joint and secured by sutures.
  Interventions: Other: Tissue Engineered Product
- N-CAM (tissue engineered product) (Experimental): N-Cell activated Matrix (CAM) is based on autologous nasal chondrocytes expanded and further cultured on type I/III collagen membrane for 2 days only to allow the cells to adhere. The IMP is implanted in the knee joint and secured by sutures.
  Interventions: Other: Tissue Engineered Product

INTERVENTIONS:
Other: Tissue Engineered Product — Implantation of tissue engineered products
  Other Names: N-TEC (tissue); N-CAM (Cell activated matrix)

SUMMARY:
The purpose of this study is to investigate the efficacy of an engineered cartilage transplant (N-TEC) in comparison to a cell-activated matrix (N-CAM) for the treatment of articular cartilage lesions in the knee. The main innovations in this trial are the use of nasal chondrocytes and the implantation of a tissue in contrast to cells seeded on a matrix. The goals of the trial are to: (i) evaluate whether implantation of a more mature graft (tissue therapy) is beneficial for the quality and durability of the repair tissue and the clinical outcome, (ii)determine the potential of the mature graft to integrate with the adjacent cartilage and form hyaline repair tissue and (iii) assess the efficacy of each treatment in correlation to the characteristics of the defect (e.g. "acute" versus "chronic" setting).

DETAILED DESCRIPTION:
Although cartilage damages in the joint develop mostly in older people due to degeneration of the cartilage, they also occur regularly in young people due to accidents. Especially in large cartilage defects there is no spontaneous self-healing. If these defects are left untreated, the risk of the development of osteoarthritis later on is significantly increased. However, the current treatment options for these defects involve difficult operation techniques, require tedious rehabilitation and are limited in the application for large injuries and the availability/quality of the donor material. Furthermore, they often lead to not entirely satisfactory clinical results due to the low quality of the repair tissue. In many cases permanent pain and restricted mobility persist. Even the use of the new cell therapies has not led to satisfactory results in the long term. An innovative promising approach is tissue engineering, where cartilage is manufactured in the laboratory using the body's own cells. First results of a clinical phase I study show that the use of engineered nasal cartilage for the regeneration of articular cartilage (knee joint) is feasible and safe. In addition the preliminary clinical results regarding the efficacy are also promising.

The goal of this phase II clinical study is to compare the efficacy of the tissue therapy with the one of the cell therapy. In order to achieve this the investigators will enroll 108 patients in the study and divide them in two groups, one receiving the cell therapy and the other the tissue therapy. Patients must display a symptomatic, isolated cartilage lesion grade III-IV (according to the grading by the International Cartilage Repair Society (ICRS)) from 2 to 8 cm2 on the femoral condyle and/or the trochlea, have to be between 18-65 years old and must consent in oral and written manner in order to be enrolled in the study. After written informed consent has been obtained, the patients will be tested to see if they comply with all other inclusion and exclusion criteria. Subsequently blood (72ml) and a cartilage biopsy (tissue sample) from the nasal septum of the patient will be taken. The cartilage cells (Chondrocytes) are isolated from the tissue, expanded for 2 weeks and placed on a collagen matrix. For the cell therapy the resulting construct will be cultured for 2 more days to allow the cells to adhere to the matrix. For the tissue therapy the construct will be cultured for 2 more weeks, to allow the cells to form cartilage tissue. After performing the quality tests the implant will be released by the manufacturer based on the sterility, cell viability and in case of the tissue therapy product the deposition of matrix. Subsequently, the construct will be implanted in the knee. At 6 weeks as well as 3, 12 and 24 months after the operation follow-ups will be performed. During the follow-ups at 12 and 24 months questionnaires (KOOS, Euro Quality of Life (EQ)-5d) will be filled out by the patient and MRIs will be performed at 3,12 and 24 months.

While the questionnaires (especially the Knee injury and Osteoarthritis Outcome Score (KOOS-Score)) provide subjective information about the efficacy of the treatment, the MRIs will shed light on the integration of the implant in the defect and give information about the quality of the repair tissue. Retrospectively the data will be analyzed in correlation to the status of the defect at time of treatment: acute (symptoms since less than 2 years) or chronic (symptoms since more than 2 years). This will give an indication whether one treatment (cell or tissue therapy) is more effective for a defined indication (acute or chronic) than the other.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥18 and ≤65 years old at time of screening.

  * Patient has a localized articular cartilage defect of the femoral condyle and/or the trochlea of the knee. 2 localized cartilage defects are accepted if the total defect size is ≤ 8 cm2, both cartilage defects are located at the femoral condyle and/or the trochlea and both cartilage defects are to be treated with N-CAM or N-TEC.
  * Patient has a defect of grade 3 or 4 according to the ICRS classification.
  * Patient has a defect size ≥2 and ≤8 cm2 as assessed by MRI/arthroscopy.
  * Patient has an intact (≤ICRS Grade 2 ) articulating joint surface (no "kissing lesions").
  * Patient has an intact meniscus (maximum 1/2-resection).
  * Patient has a stable knee joint or sufficiently reconstructed ligaments. If not, ligament repair has to be done during the operation or within 6 weeks of the planned cartilage treatment.
  * Patient has a maximum baseline score of 75/100 in the KOOS subjective knee evaluation.
  * Patient is willing and able to give written informed consent to participate in the study and to comply with all study requirements, including attending all follow-up visits and assessments and to complete postoperative rehabilitation regimen.

Exclusion Criteria:

* Patient is the investigator or any sub-investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol or in a dependency or employment with the sponsor.
* Patient is unable to understand the patient information
* Patient is unable to undergo magnetic resonance imaging (MRI) or is sensitive to gadolinium
* Patient has had prior surgical treatment of the target knee within 12 months using mosaicplasty and/or microfracture (Note: prior diagnostic arthroscopy with debridement and lavage are acceptable within 12 months). Anterior cruciate ligament repair is accepted, if the target knee is stable or a primary Anterior cruciate ligament (ACL) reconstruction is performed within 6 weeks of the planned cartilage treatment.
* Patient has a relevant meniscus tear. Partial meniscal removal allowed, if not exceeding 1/2. Meniscus suture is not allowed in parallel, but if successful, cartilage treatment might be added 12 months later.
* Patient has radiologically apparent degenerative joint disease in the target knee as determined by Kellgren and Lawrence grade >2.
* Patient has chronic inflammatory arthritis, and/or infectious arthritis.
* Patient has an unstable knee joint or insufficiently reconstructed ligaments. If ligament repair is necessary, the repair has to be performed during the operation or within 6 weeks of the planned cartilage treatment.
* Patient has malalignment (no valgus- or varus-deformity) in the target knee ≥ 5°. In suspected cases, the mechanical axis must be established radiographically through complete leg imaging during standing and in a.p. or rather p.a. projection. If alignment surgery is necessary, surgery has to be performed within 6 weeks of the planned cartilage treatment.
* Patient has an osteochondral defect (defined as bony substance defect of >3mm depth). Bone marrow edema is allowed.
* Patient has relevant bilateral lower limb pain.
* Patient has a known systemic connective tissue disease.
* Patient has a known autoimmune disease.
* Patient has a known immunological suppressive disorder or is taking immunosuppressives.
* Patient is currently systemically or intra-articularly taking steroids and/or has used steroids within the 30 days prior to the planned treatment.
* The patient has a known history of HIV/AIDS. (Protection of staff)
* The patient has a known history of Treponema pallidum (syphilis). (Protection of staff)
* The patient has an active hepatitis B or C infection with verified antigens. Patients with a cured hepatitis B or C infection and/or verified antibodies are not excluded. (Protection of staff)
* The patient has at the site of surgery an active systemic or local microbial infection, eczematization or inflammable skin alterations (including protozoosis: Babesiosis, Trypanosomiasis (e.g. Chagas-Disease), Leishmaniasis, persistent bacterial infections, such as Brucellosis, spotted and typhus fever, other Rickettsiosis, Leprosy, Recurrent Fever, Melioidosis or Tularaemia).
* Patient has a known history of cancer.
* Patient has a known history of primary hyperparathyroidism, hyperthyroidism, reduced kidney function, chronic renal failure or prior pathological fractures, independent of the genesis.
* Patient has any degenerative muscular or neurological condition that would interfere with evaluation of outcome measures including but not limited to Parkinson's disease, amyotrophic lateral sclerosis (ALS), or multiple sclerosis (MS).
* Patient has a body mass index (BMI) >35 kg/m2.
* Patient is pregnant, lactating or anticipates becoming pregnant within 24 months after surgery.
* Patient is currently participating, or has participated in any other clinical study within 3 months prior to the screening visit.
* Patient has known current or recent history of illicit drug or alcohol abuse or dependence defined as the continued use of alcohol or drugs despite the development of social, legal or health problems.
* Patient has psychiatric or cognitive impairment that, in the opinion of the investigator, would interfere with the patient's ability to comply with the study requirements, e.g., Alzheimer's disease.
* Patient has any other condition, which, in the opinion of the investigator, would make the patient unsuitable for the study.
* Patient is unable to tolerate local anesthesia
* Any known allergies, especially for porcine collagen, penicillin or streptomycin
* Patient is unwilling and/or unable to give written informed consent to participate in the study and to comply with all study requirements, including attending all follow-up visits and assessments and to complete postoperative rehabilitation regimen.

Intraoperative Exclusion Criteria:

* Patient has a total defect size <2 or defect size extends graft size and could therefore not be treated in total.
* Patient has >2 independent cartilage lesions
* Patient has symptomatic full-thickness (ICRS Grade 3 or 4) of patella or tibial plateau.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
comparison of the efficacy of the two investigational medicinal products (IMPs) | 24 months
  Assessment whether a tissue therapy will improve the clinical efficacy for the patient, leading to an increase of at least 10 points in the main primary outcome (self-assessed score KOOS) after 24 months as compared to the cell therapy group

SECONDARY OUTCOMES:
stability and Integration of the implanted IMP | 24 months
  Assessment of the stability and Integration of the graft with the adjacent tissues by magnetic resonance observation of cartilage repair tissue (MOCART Score) derived from the MRI as well as the remodeling of the implanted grafts towards native cartilage assessed by delayed gadolinium-enhanced MRI of cartilage (dGEMRIC) evaluation from the 24-month follow-up
efficacy for patient | 24 months
  Improvement of the KOOS-Score from baseline to 24 months

OTHER OUTCOMES:
efficacy of IMPs related to acute vs. chronic lesions | 24 months
  Determination if one treatment is more beneficial than the other in a certain setting (onset of symptoms) (retrospective Analysis)
safety of IMPs | 24 months
  Assessment of number of serious adverse drug reaction (SADRs) or suspected unsuspected serious adverse reaction (SUSARs)

CONTACTS AND LOCATIONS:
Overall Officials: Marcel Jakob, Prof. Dr., Study Chair — University Hospital, Basel, Switzerland
Locations (5):
- University Hospital Sveti Duh, Zagreb, Croatia
- Germany (2):
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Orthopädische Klinik König-Ludwig-Haus, Würzburg
- Istituto Ortopedico Galeazzi (IOG), Milan, Italy
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mumme M, Wixmerten A, Ivkovic A, Peretti GM, Yilmaz T, Reppenhagen S, Pullig O, Miot S, Izadpanah K, Jakob M, Mangiavini L, Sosio C, Vuletic F, Bieri O, Biguzzi S, Gahl B, Lehoczky G, Vukojevic R, Hausner S, Gryadunova A, Haug M, Barbero A, Martin I. Clinical relevance of engineered cartilage maturation in a randomized multicenter trial for articular cartilage repair. Sci Transl Med. 2025 Mar 5;17(788):eads0848. doi: 10.1126/scitranslmed.ads0848. Epub 2025 Mar 5. PMID 40043142

DOCUMENTS (2):
  • Study Protocol (2018-04-10): https://cdn.clinicaltrials.gov/large-docs/05/NCT02673905/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-28): https://cdn.clinicaltrials.gov/large-docs/05/NCT02673905/SAP_001.pdf